CLINICAL TRIAL: NCT05512143
Title: Targeting the Brain-heart Axis With TMS Among Reproductive Aged Women With PTSD
Brief Title: TMS for PTSD and Blood Pressure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Margaret Bublitz, Staff Psychologist, Lifespan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1952743
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Post-traumatic Stress Disorder; Hypertension
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Hypertension | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TMS (Experimental): Participants will receive active TMS to the left dorsolateral prefrontal cortex (DLPFC). Right DLPFC will be targeted using a modification of the Beam method. TMS will be administered at 10Hz, 120% of motor threshold, 3000 pulses per session
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Participants will undergo a standard course of TMS treatment (30 sessions/6 weeks).

SUMMARY:
In this randomized clinical trial, we will test the short and longer term effects of repetitive transcranial magnetic stimulation (TMS) on blood pressure among reproductive aged female participants with elevated symptoms of post-traumatic stress disorder and hypertension.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death and disability for women in the United States. Posttraumatic Stress Disorder (PTSD) affects 1 in 20 reproductive aged women and significantly increases risk CVD. In the perinatal period, cardiovascular complications account for one third of maternal deaths, and emerging evidence indicates that PTSD increases risk for pregnancy-related CVD. As well, exposure to cardiovascular complications in pregnancy increases risk for CVD later in life. Therefore, effective treatment of PTSD in reproductive aged women, prior to disease, holds significant potential to decrease risk for CVD onset across the life course. Repetitive transcranial magnetic stimulation (TMS) is a safe, non-invasive, promising novel approach to treat PTSD and reduce risk for CVD. TMS dramatically reduces PTSD symptoms, and a single session of non-invasive brain stimulation methods, including TMS, reduce heart rate and blood pressure, and increase heart rate variability. However, lack of knowledge on the long-term autonomic benefits of TMS prevents utilization of this intervention for patients at risk for CVD. In this COBRE Center for Neuromodulation pilot study, we aim to determine the acute and longer-term effects of TMS on blood pressure in women at risk for CVD. We propose a single arm trial of TMS among 20 women with elevated PTSD symptoms who also have a diagnosis of hypertension. All participants will receive active TMS to the left dorsolateral prefrontal cortex (DLPFC) administered at 10Hz, 120% of motor threshold, 3000 pulses per session. At the first TMS session, blood pressure, heart rate, and heart rate variability will be monitored for 20 minutes before, during, and after TMS to evaluate acute cardiovascular changes to TMS. Throughout the intervention and at 1-month post intervention, participants will complete 24-hour blood pressure monitoring and PTSD symptom assessments to enable examination of longer-term effects of TMS on blood pressure, as well as test the temporal associations between change in PTSD symptoms and blood pressure. The specific aims of the study are to: examine change in 24-hour blood pressure following a standard course of TMS (Aim 1), and examine if change in PTSD symptoms is associated with changes in 24-hour blood pressure among reproductive aged women with elevated PTSD symptoms (Aim 2). The current proposal is closely aligned with the research priorities described by the NHBLI working group on hypertension to 1) support clinical trials for early intervention for high blood pressure, particularly in younger populations, and 2) support studies related to the role of sex differences in the complications of hypertension and hypertension in pregnancy. Results from this pilot project will establish a new line of inquiry in neuromodulation for PI Bublitz and will provide essential pilot data for a future R01 application to conduct a mechanistic sham-controlled clinical trial of TMS for treatment of PTSD and hypertension in at-risk women.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, 18-44 years old, PCL-5 score of > 31 at enrollment or PHQ2 > 3 at enrollment, physician-diagnosed hypertension, in stable psychiatric treatment

Exclusion Criteria:

* pregnant; active suicidality or psychosis; bipolar I disorder; a seizure disorder and/or seizure disorder in a first degree relative; any metal in the skull; greater than moderate substance use disorder (except nicotine or cannabis) in the prior 6 months

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 6 weeks
  Change in 24-hour blood pressure before and after TMS intervention

SECONDARY OUTCOMES:
PTSD symptoms | 6 weeks
  Change in PTSD symptoms from baseline to follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Lifespan Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No